CLINICAL TRIAL: NCT00046202
Title: Investigations Into Inborn Errors of Cholesterol Synthesis and Related Disorders
Brief Title: Study of Inborn Errors of Cholesterol Synthesis and Related Disorders
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020311; 02-CH-0311
Record Dates: First submitted 2002-09-21; First posted 2002-09-23 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-09-26

CONDITIONS: Lysosomal Storage Disease; Cholesterol Metabolism
Keywords: Inborn Error of Cholesterol Synthesis; Cholesterol; Lysosomal Storage; Natural History; Inborn Errors of Cholesterol Synthesis; Smith-Lemli-Optiz Syndrome; Lathosterolosis; Desmosterols; CHILD Syndrome; Greenberg Dysplasia; X Linked Dominant Chrondrodysplasia
MeSH Terms: conditions — Lysosomal Storage Diseases; Lathosterolosis; Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects; HEM dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal subjects: subjects in whom no disorder of cholesterol is suspected related to affected individuals
- subjects suspected of cholesterol disorder: subjects in whom a disorder of cholesterol metabolism is suspected

SUMMARY:
This study will investigate the cause and medical problems associated with a group of genetic disorders known as inborn errors of cholesterol synthesis, in which the body does not produce cholesterol. People with this disorder may have birth defects and learning and behavioral problems.

People with an inborn error of cholesterol synthesis and related disorders, including Smith-Lemli-Opitz syndrome, lathosterolosis, desmosterolosis, X-linked dominant chondrodysplasia, CHILD syndrome, Greenberg dysplasia, and some cases of Antley-Bixler syndrome, may be eligible for this study. People who are carriers of the disorders also may enroll.

Participants and family members will provide blood and urine samples, as well as other tissue samples collected during medically indicated procedures such as biopsy or surgery. These tissues may include, for example, gallstones, cataracts, cerebrospinal fluid, amniotic fluid, lymph tissue, and DNA samples. In rare instances, a skin biopsy may be requested to aid in establishing a diagnosis.

Medical information will also be gathered from medical records, photographs, and X-rays.

DETAILED DESCRIPTION:
It is known that inborn errors of cholesterol synthesis give rise to human malformation/cognitive impairment syndromes. Smith-Lemli-Opitz syndrome is the prototypical example of a post-squalene inborn error of metabolism; however, this group of disorders now includes lathosterolosis, desmosterolosis, X-linked dominant chondrodysplasia (CDPX2), CHILD syndrome, HEM dysplasia, and some cases of Antley-Bixler syndrome (1-3). Due to the extremely rare occurrence of some of these disorders, the full phenotypic spectrum has yet to be defined. Cholesterol transport in cells can also cause a disorder known as Niemann-Pick Disease type C (NPC). NPC belongs to a group of disorders known as lysosomal storage disorders. The purpose of this protocol is to 1) allow for the collection of biomaterial and medical information that can be studied to gain insight into the pathological processes; 2) allow for the collection of DNA and medical information from individuals who have a phenotypic resemblance to known disorders of cholesterol synthesis, lysosomal storage disorders or individuals who may be carriers of these disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be eligible for this study if they have or are suspected to have an inborn error of cholesterol synthesis or if they are related to a proband with a suspected inborn error of cholesterol synthesis. No exclusions will be made based on gender, ethnicity or age.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Convenience sampling: affected patients and their relatives, samples from biorepositories
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2002-10-09 (Actual)

PRIMARY OUTCOMES:
sample collection | event driven upon enrollment
  collect sample to study rare manifestations or disease

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared in aggregate related to the disorders represented by accrual.

REFERENCES:
- [Background] Kelley RI, Hennekam RC. The Smith-Lemli-Opitz syndrome. J Med Genet. 2000 May;37(5):321-35. doi: 10.1136/jmg.37.5.321. PMID 10807690
- [Background] Nwokoro NA, Wassif CA, Porter FD. Genetic disorders of cholesterol biosynthesis in mice and humans. Mol Genet Metab. 2001 Sep-Oct;74(1-2):105-19. doi: 10.1006/mgme.2001.3226. PMID 11592808
- [Background] Kelley RI, Kratz LE, Glaser RL, Netzloff ML, Wolf LM, Jabs EW. Abnormal sterol metabolism in a patient with Antley-Bixler syndrome and ambiguous genitalia. Am J Med Genet. 2002 Jun 15;110(2):95-102. doi: 10.1002/ajmg.10510. PMID 12116245
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-CH-0311.html